CLINICAL TRIAL: NCT02642588
Title: Effect of a Commercially Available Carbohydrate Rich Gel on Maternal Fatigue: A Randomized Controlled Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Melissa March (Unknown); Alison Bauer (Unknown); Gaetan Pettigrew (Unknown); Daisy Hassani (Unknown); Celina Cunanan (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UHCaseMC
Record Dates: First submitted 2015-12-24; First posted 2015-12-30 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Effect of Carbohydrate Ingestion During Active Labor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- energy gel (Experimental): women will be given 22 g of carbohydrates every 45-60 minutes for up to 8 hours or until delivery during the active phase of labor
  Interventions: Dietary Supplement: energy gel
- control (No Intervention): women will be given only clear liquids during labor

INTERVENTIONS:
Dietary Supplement: energy gel — energy gel: gelatinous edible containing carbohydrates typically used during endurance races
  Arms: energy gel

SUMMARY:
Women in active labor will be given energy gel at 45-60 minute intervals and their fatigue level will be compared to women receiving usual practice care i.e. clear liquids only.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or older as well as willing and able to provide informed consent
* Patients with BMI < 35 kg/m^2
* Gestational age >37 weeks

Exclusion Criteria:

* - Patients younger than 18 years,
* Patients unable or unwilling to provide informed consent,
* Patients who are illiterate,
* Patients who are non-English speaking or reading,
* Patients who are University Hospital employees,
* Patients undergoing induction of labor for maternal or fetal indications other than elective induction after 39 weeks or induction for post-term pregnancy
* Multi-fetal gestations (>1 intrauterine pregnancy),
* Patients with a history of GI disorders such as hyperemesis gravidarum, inflammatory bowel disease or irritable bowel syndrome
* Patients with an increased risk of aspiration such as BMI >35 kg/m^2, severe GERD, gastroesophageal motility disorders,
* Patients with acute or chronic platelet dysfunction (e.g.: idiopathic thrombocytopenic purpura, HELLP syndrome) which may necessitate need for general anesthetic for Cesarean delivery
* Patients with history of peptic ulcer disease,
* Patients who have a contraindication to epidural placement and would require general anesthestetic in event of Cesarean delivery
* Patients with suspected or proven placenta accreta, increta or percreta,
* Patients with excessive nausea or vomiting during labor
* Patients with a history of food allergies or allergies to specific components found in the energy gel.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2018-02 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue | every 2 hours until delivery
  evaluated by visual analog scale
duration of labor | from start of active phase until delivery
  will measure time to delivery and duration of 2nd stage of labor